CLINICAL TRIAL: NCT02330861
Title: Relationship Between Pressure and Flow Velocity on Coronary Physiology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Kenichi Fujii, Relationship between pressure and flow velocity on coronary physiology, Hyogo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KFujii-000000
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2017-02

CONDITIONS: Coronary Stenosis
Keywords: Coronary Circulation
MeSH Terms: conditions — Coronary Stenosis

ARMS (1):
- Normal coronary artery (Other)
  Interventions: Device: combowire and IVUS

INTERVENTIONS:
Device: combowire and IVUS

SUMMARY:
Subjects are patients who are planned to do percutaneous coronary intervention for coronary stenosis in the left circumflex artery without other stenosis in the left ascending artery and the right coronary artery, or a patient with normal coronary artery. Immediately after coronary angiography or percutaneous coronary intervention, the investigators will evaluate for coronary hemodynamics by distribution of wave intensity which is calcurated by coronary pressure and flow velocity with Combowire in each coronary segment. Also, they will assess coronary morphology by View It in each coronary segment.

DETAILED DESCRIPTION:
Combowire (Volcano Therapeutics Inc., CA, USA) is a 0.014 inch pressure/Doppler sensor-tipped-guidewire which can measure coronary pressure and flow velocity.

View It (Terumo Co., Japan) is a guide catheter with intravascular ultrasound which can measure coronary morphology such as vessel diamter.

ELIGIBILITY:
Inclusion Criteria:

* A patient who are planned to do percutaneous coronary intervention for stenosis in the left circumflex artery without any lesions in other coronary arteries
* Or a patient who is performed coronary angiography without significant stenosis lesion in 3-coronary vessel

Exclusion Criteria:

* A patient with coronary stenosis with LAD
* Hemodialysis
* Acute coronary syndrome
* Congestive heart failure
* A patient with shock vitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Wave intensity | Immediately after coronary angiography or percutaneous coronary intervention

SECONDARY OUTCOMES:
Coronary pressure | Immediately after coronary angiography or percutaneous coronary intervention
Flow velocity | Immediately after coronary angiography or percutaneous coronary intervention
Vessel diameter | Immediately after coronary angiography or percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hyogo College of Medicine, Nishinomiya, Japan